CLINICAL TRIAL: NCT06393465
Title: Real-World Effectiveness of High-Dose Tafamidis on Neurologic Disease Progression in Mixed-Phenotype Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Brief Title: Real-World Effectiveness of High-Dose Tafamidis on Neurologic Disease Progression in Mixed-Phenotype Transthyretin Amyloid Cardiomyopathy
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461121; NCT06393465 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Transthyretin Amyloidosis Cardiomyopathy (ATTR-CM)
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mixed phenotype ATTR-CM: ATTR-CM patients presenting with mixed phenotype
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 61 milligrams under real world conditions
  Other Names: Vyndamax

SUMMARY:
This study will examine the clinical effectiveness of Tafamidis in patients with Mixed Phenotype Transthyretin Amyloidosis using data that already exist in patients' medical records

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at diagnosis.
* Diagnosed with ATTRv-CM or ATTRwt-CM, mixed phenotype.
* Treated with tafamidis, as VYNDAMAX 61 mg (one 61-mg tafamidis capsule) orally once daily for ≥12 months or started on tafamidis 20 mg then switched to VYNDAMAX 61 mg for ≥12 months
* Have had ≥1 pre- and ≥1 post-treatment neurologic assessments.

Exclusion Criteria:

* History of any organ transplant.
* Individuals who are non-ambulatory.
* Prior or current treatment with any disease-modifying therapy (investigational or approved) alone or in combination, except tafamidis, as VYNDAQEL 80 mg [four 20-mg tafamidis meglumine capsules] orally once daily or VYNDAMAX 61 mg [one 61-mg tafamidis capsule] orally once daily.
* Peripheral neuropathy attributed to causes other than ATTR amyloidosis (eg, diabetes mellitus, B12 deficiency, hypothyroidism, shingles,Lyme disease, HIV infection, secondary to injury, chronic kidney disease).
* Patient's data fails to pass data quality checks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with mixed-phenotype ATTR-CM who are treated in the Amyloidosis Program at MedStar in the U.S and three other study sites (Canada, Portugal and Italy).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Rate of neurologic disease progression | Baseline through at least 12 months of treatment
  Describe and compare the rate of neurologic disease progression before and after initiation of tafamidis in patients with mixed-phenotype ATTR-CM receiving tafamidis 61 mg daily in a real world setting.

SECONDARY OUTCOMES:
Change from Baseline in modified Body Mass Index (BMI) | Baseline (BL) through at least 12 months of treatment
  Assess change from BL in mBMI in patients with mixed phenotype ATTR-CM 61 mg tafamidis

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461121